CLINICAL TRIAL: NCT05952947
Title: A Multicenter, Single Arm, Open Label, Phase I Clinical Study to Evaluate the Safety, Tolerability and Efficacy of HRYZ-T101 Injection for HPV18 Positive Solid Tumor
Brief Title: HRYZ-T101 Injection for HPV18 Positive Solid Tumor
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: HRYZ Biotech Co. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-T01-C2001
Record Dates: First submitted 2023-07-05; First posted 2023-07-19 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2023-06

CONDITIONS: Cervical Cancer; Head and Neck Squamous Cell Carcinoma; Carcinoma of Vagina; Carcinoma of Penis; Anal Cancer; Carcinoma of Vulva
MeSH Terms: conditions — Uterine Cervical Neoplasms; Squamous Cell Carcinoma of Head and Neck; Vaginal Neoplasms; Penile Neoplasms; Anus Neoplasms; Vulvar Neoplasms | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRYZ-T101 Injection (Experimental): Patients will undergo lymphocytapheresis, then treatment with HRYZ-T101 TCR-T cells.
  Interventions: Biological: HRYZ-T101 Injection; Drug: Fludarabine + Cyclophosphamide

INTERVENTIONS:
Biological: HRYZ-T101 Injection — On day 1, the TCR-T cells will be administered intravenously.
Drug: Fludarabine + Cyclophosphamide — Fludarabine: 25mg/m²/day×3days; Cyclophosphamide: 250mg/m²/day×3 days

SUMMARY:
A multicenter, open label, single arm dose escalation phase I study to evaluate the safety, tolerability, and efficacy of HRYZ-T101 injection for HPV18 positive solid tumor. The study will investigate RP2D of HRYZ-T101 TCR-T cell injection.

ELIGIBILITY:
Inclusion Criteria:

* 1. The patient must be willing to sign the informed consent form.
* 2. Age ≥18 years and ≤75 years.
* 3. Metastatic or recurrent solid tumors with confirmed HPV18 infection based on TNM & FIGO staged histopathological investigation. .
* 4. Subjects who have failed anti-tumor treatment in the past and lack effective treatment options.
* 5. HPV18 positive and HLA-DRB1*0901 allele.
* 6. ECOG performance status ≤1.
* 7. Estimated life expectancy ≥ 3 months.
* 8. Patients must have at least one measurable lesion defined by RECIST 1.1.
* 9. Patients with any organ dysfunction as defined below:

  1. Leukocytes≥3.0 x 10^9/L;
  2. blood platelets ≥75 x 10^9/L;
  3. hemoglobin≥85g/L;
  4. Absolute lymphocyte count≥0.8 x 10^9/L
  5. Serum albumin ≥ 30g/L;
  6. total bilirubin≤1.5×ULN; ALT/AST≤3×ULN or ≤5×ULN for liver metastases;
  7. Creatinine clearance ≥50mL/min; or serum creatinine ≤1.5×ULN;
  8. INR≤1.5×ULN; APTT≤1.5×ULN;
  9. LVEF≥50%;
  10. SpO2≥92%.
* 10. Subjects with potential fertility must agree to use effective contraceptive methods during the whole trials period and at least 1 year after receiving HRYZ-T101 cell transfusion treatment. HCG test for female with potential fertility must be negative within 7 days before apheresis.

Exclusion Criteria:

* 1. Have a history of hypersensitivity to cyclophosphamide or fludarabine, and it is known that any ingredient used in the treatment of this study will produce allergic reactions.
* 2. Those who have undergone systemic anti-tumor treatment within 4 weeks before apheresis, including who have received conventional chemotherapy, large-area radiotherapy, targeted therapy, immunotherapy or biological therapy, and other anti-tumor treatment. Have received small molecule targeted drugs and oral fluorouracils or Chinese herbal medicine within 2 weeks before apheresis.
* 3. Have received any investigational drug within 4 weeks before apheresis, or have participated in another clinical study at the same time.
* 4. Have received any cell therapy products before.
* 5. Those who have undergone major surgery within 4 weeks before apheresis, or minor surgery within 2 weeks before apheresis.
* 6. Toxicity of previous treatment has not been mitigated or ≤ Grade 1 before apheresis.
* 7. Have received live attenuated vaccine or adenovirus vector vaccine within 4 weeks before apheresis.
* 8. Have central nervous system metastasis with symptoms.
* 9. Subjects with clinical cardiac symptoms or diseases that cannot be well controlled.
* 10. Subjects with serious or uncontrolled systemic disease or any unstable systemic disease.
* 11. Subjects with active infection requiring systemic treatment with anti-infective drugs within 2 weeks before apheresis.
* 12. Subjects have any active autoimmune disease or history of autoimmune disease.
* 13. Have received immunosuppressive agents, or systemic corticosteroids, immunomodulators within 2 weeks before apheresis.
* 14. Subjects with other malignant tumors. Except for: (1) Carcinoma in situ with curative treatment and no evidence of recurrence for at least 2 years; (2) the primary malignant tumor has been completely resected and achieved CR for ≥ 2 years.
* 15. Subjects with history of thromboembolism ≥ Grade 3 within 6 months before apheresis, or is receiving thrombolytic or anticoagulant for high-risk of thromboembolism.
* 16. Known HIV or syphilis infection, and/or active hepatitis B virus or hepatitis C virus infection.
* 17. Organ transplanters and allogeneic cell transplanters.
* 18. Subjects with active pulmonary tuberculosis infection within 1 year or have not received treatment at least 1 year before apheresis.
* 19. Pregnant or lactating female, or those whose HCG test is positive before enrollment.
* 20. According to the judgment of the researcher, those who are not suitable for the group, such as poor compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
DLT | 28 days
  Dose-limiting toxicity
Adverse events and serious adverse events | 2 years
  Incidence of adverse events and serious adverse events

SECONDARY OUTCOMES:
Objective Response Rate（ORR） | 2 years
  The percentage of subjects with PR or CR assessed by RECIST 1.1.
Disease Control Rate (DCR) | 2 years
  The percentage of subjects with a confirmed CR, PR, or stable disease (SD) assessed by RECIST 1.1.
Duration of response (DoR) | 2 years
  Subjects who show a confirmed CR or PR as assessed by RECIST 1.1.
Time to response (TTR) | 2 years
  Time from date of T-cell administration to first documented evidence of confirmed (CR or PR) as assessed by RECIST 1.1.
Progression-Free Survival（PFS） | 2 years
  The length of time from enrollment until the time of progression of disease.
Overall Survival (OS) | 2 years
  The interval of time between the date of T-cell infusion and the date of death.
Duration of TCR T cells in-vivo persistence | 2 years
  Blood samples were collected to measure persistence of infused HRYZ-T101.
Concentration of Cytokines (IL-2、IL-6、IL-10、TNFα、IFNγ) | 2 years
  Collect blood samples and analyze for presence of cytokines (IL-2、IL-6、IL-10、TNFα、IFNγ) at specified intervals before and after treatment with HRYZ-T101.

OTHER OUTCOMES:
Number of Subjects with positive anti-drug antibodies (ADA) | 2 years
  Serum samples will be collected to analyze for the presence of ADAs using validated immunoassays.
Number of subjects with replication competent lentivirus (RCL) | 2 years
  RCL exposure will be assessed by polymerase chain reaction (PCR) based assay.
T cell subgroup in peripheral blood | 2 years
  Collect blood samples and analyze for T cell subgroup by flow cytometry at specified intervals before and after treatment with HRYZ-T101.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua Wu, Doctor, Principal Investigator — Fudan University; Jian Zhang, Doctor, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No